CLINICAL TRIAL: NCT01303302
Title: The TANTALUS® II for the Treatment of Type 2 Diabetes: A Single-Blind Cross-Over Study
Brief Title: The TANTALUS® II for the Treatment of Type 2 Diabetes
Acronym: Crossover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaCure (USA), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MC CP TAN2007-032; Cross-over (Other: MetaCure (USA))
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: C19 246 300
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GCM stimulation (Active Comparator): The patient will be implanted with a gastric contractility modulation (GCM) stimulation system using the TANTALUS System for treatment of type 2 diabetic patients.
  Interventions: Device: Tantalus System
- Device off (Sham Comparator): The TANTALUS System is implanted but is off
  Interventions: Device: TANTALUS system

INTERVENTIONS:
Device: Tantalus System — The TANTALUS System is an active implantable device, generating Gastric contractility modulation (GCM) stimulation for the treatmnet of type 2 diabetes
  Other Names: TANTALUS II
  Arms: GCM stimulation
Device: TANTALUS system — The TANTALUS System is an active implantable device, generating Gastric contractility modulation (GCM) stimulation for the treatmnet of type 2 diabetes. In the sham comparator the device is off.
  Other Names: TANTALUS II
  Arms: Device off

SUMMARY:
Evaluation of the safety and efficacy of gastric contractility modulation (GCM) stimulation using the TANTALUS System in the improvement of glycemic control measured by changes in HbA1c. Effects of GCM on weight loss and associated co-morbid conditions will also be evaluated

DETAILED DESCRIPTION:
This is a multi-center, single blind, randomized, cross-over study. Subject enrollment will continue until forty (40) eligible participants have been randomized into one of the two groups. Subjects will undergo baseline valuation (Visit 1) during which the stability of their glycemic parameters, medical treatment and medical condition will be assessed. Subjects meeting all inclusion/exclusion criteria at Visit 2 will be implanted. Approximately three days prior to their implantation, subjects will be seen for their 'pre-implant' medical evaluation (Visit 3). One week after implant (Visit 5, Week 1)subjects will be randomized into one of two groups (A and B).

"Group A" subjects will have their device programmed to deliver GCM signal including the setting of automatic eating detection parameters for the first 24 week period (Period 1). At Visit 10, (week 25 and end of Period 1), Group A subjects will have their devices turned "OFF" for the next 24 weeks period (Period 2). At Visit 15, (week 49 and end of Period 2), Group A subjects will have their devices turned "On" for the next 24 weeks period (Period 3) "Group B" subjects will not have their device activated for the first 24 weeks (Period 1) of their study. At Visit 10 (week 25 end of Period 1), Group B subjects devices will have their device turned "ON" (i.e. activated to deliver CGM signals) for the 24 weeks period (Period 2). At Visit 15, (week 49 and end of Period 2), Group B subjects will have their devices turned "OFF" for the next 24 weeks period (Period 3).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 through 70 years of age
* Body mass index >=28 and <=45 (kg/m2)
* Type 2 diabetes duration more than 6 month
* Type 2 diabetic sublecys treated with oral anti-diabetic agents
* Stable anti-diabetic medication for at least 3 month prior to enrollment
* HbA1c >=7.5% and <=9.5% on visit 1; subjects with T2DM duration .10 years should have <=9.0% at visit 1
* Stable HbA1c, defined as no significant change (variation <=0.5%)between a historical value recorded in the subject's medical record with in 3 month prior to enrollment and the HbA1c gathered at visit 1
* Fasting blood glucose >120 and < 240 mg/dl on visit 1; subjects with T2DM duration > 10 yaers should have .120 ans<=180 mg/dl at visit 1
* Women with child bearing potential (i.e, not post menopausal or surgically sterilized) must agree to use adequate birth control methods
* Stable weight, defined as no significant weight change (variation <5%)within three months prior to enrollment
* If taking these medication, stable anti-hepertensive and lipid-lpwering medication for at least one month prior to enrollment
* If subject is under unti-depressant medication the treatment needs to be stable for at least six month prior to enrollment
* Wllingness to refrain from using prescription, over the counter or herbal weight loss product for the duration of the trial
* Ability and willingliness to perform required study and data collection procedures and adhere to operating requirements of the TANTALUS II Syatem
* Alert, mentally competant, and able to understand and willing to comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial
* Able to provide voluntary informed consent

Exclusion Criteria:

* Insulin therapy
* Taking GLP-1 analogue, such as exenatide (Byette) in the last 3 month before enrollment Taking medication known to affec gastric mobility such as narcotics (chronic use) and anticholinergics/antispasmodics
* Use of prescription, over the counter or herbal weight loss product or obesity drugs during the past two month
* Experiencing sever and progressing diabetic complications (i.e retinopathy not stabilized, nephropathy with macroalbuminuria)
* Prior wound healing problems
* Diagnosed with past or present psychiatric condition that may impair his or her ability to comply with the study procedure
* Use of anti-pchichotic medication
* Diagnosed with an eating disorder such as bulimia or binge eating
* Obesity due to endocrinopathy (e.g.Cushing disease, Hypothyroidism)
* Hiatal hernia requiring surgical repair or paraesophageal hernia
* Pregnant or lactating Diagnosed with impared liver function (liver enzyms 3 times graeted than normal)
* Any prior bariatric surgery
* Ant history of pancreattitis Any history of peptic ulcer disease within 5 years of enrollemnt Diagnosed with gastroparesis or GI mobility disorder Use of active medical device (either implantable or external) such as ICD, pacemaker, drug infusion device, or neurostimulator (either implantable or worn) Subject using an external active device who are able anf willing to avoid use of the device during the study may be enrolled.
* Cardiac history that physician feels should exclude the subject from the study.
* Use of anotherc investigational device agent in the 30 dayes prior to enrollemnt
* A history of life threatening diseas within 5 years of enrollment
* Change in diabetic medication from between visit 1 and visit 3
* Any additional condition(S) that in the investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the differences in HbA1c levels | One year
  Comparison of the differences in HbA1c levels between treatment and control groups between changes occurred during period 2 to period 3

SECONDARY OUTCOMES:
Improvement in weigth and metabolic parameters | One year
  * Trends in weight loss will be of a reduction in weight during periods 2 and 3.
  * Trends in improvement in metabolic parameters such as waist circumference, blood pressure and lipids occurred during period 2 to period 3.
  * Difference in device related Adverse Events between treatment and control groups between periods of active and inactive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Walid Hadda, PhD, Study Director — MetaCure Limited
Locations (7):
- Medical University of Vienna, Vienna, Austria
- Germany (4):
  - Gemeinschaftspraxis Drs. Klausmann, Aschaffenburg
  - Arzt für Innere Medizin und Endokrinologie, Bad Nauheim
  - Krankenhaus Sachsenhausen, Frankfurt
  - Diabetes-Praxis Muenster, Münster
- Università Cattolica S. Cuore, Rome, Italy
- CMKP- Centrum Medyczne Kształcenia Podyplomowego, Warsaw, Poland